CLINICAL TRIAL: NCT04388371
Title: Glutamine PET Imaging in LAM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The LAM Foundation (Other)
Responsible Party: Principal Investigator, Timothy Blackwell, Principal Investigator, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 190481
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Lymphangioleiomyomatosis (LAM)
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Glutamine

STUDY DESIGN:
Intervention Model Description: Test subjects with spontaneous or tuberous sclerosis complex associated lymphangioleiomyomatosis (LAM) who have not been started on therapy with mTOR inhibitors such as sirolimus or everolimus to undergo a PET/CT scan using an novel PET tracer that may better evaluate disease activity in LAM subjects both before and after the initiation of mTOR inhibitor therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prior to subject taking sirolimus or everolimus (Experimental): To compare images from subjects prior to use of sirolimus or everolimus to images produced after use of sirolimus or everolimus.
  Interventions: Drug: Glutamine
- subjects taking sirolimus or everolimus (Experimental): To compare images from subjects prior to use of sirolimus or everolimus to images produced after use of sirolimus or everolimus.
  Interventions: Drug: Glutamine

INTERVENTIONS:
Drug: Glutamine — Glutamine will be administered by IV injection prior to PET imaging.

SUMMARY:
In this study, subjects with spontaneous or tuberous sclerosis complex associated lymphangioleiomyomatosis (LAM) who have not been started on therapy with mTOR inhibitors such as sirolimus or everolimus to undergo a PET/CT scan using an novel PET tracer that may better evaluate disease activity in LAM subjects both before and after the initiation of mTOR inhibitor therapy will be enrolled. The procedure for each scan will be similar, involving one administration of the novel tracer C11-glutamine followed by a whole body PET/CT scan.

DETAILED DESCRIPTION:
Objectives This is a hypothesis-driven prospective pilot study of the targeted PET reagent 11C-Glutamine in LAM.

The objective is to test the hypothesis that 11C-Glutamine PET/CT will demonstrate uptake within the lungs and/or associated neoplasm of patients with LAM and that this effect will be modified by treatment with mTOR inhibitors.

Rationale Our rationale is that 11C-Glutamine PET/CT may provide an improved ability to diagnose LAM, as well as predict and monitor treatment response to mTOR inhibitors.

Aims Test the hypothesis that 11C-Gln PET imaging of the lungs in humans will reflect the known "glutamine addiction" seen in mechanistic preclinical studies of LAM. As a result, PET imaging will show increased tracer uptake in affected areas of diseased lungs and will show reduced uptake after initiating treatment with mTOR inhibitors.

Approach: We will evaluate 11C-Glutamine PET/CT uptake in patients with known LAM, and if possible, we will test subjects again after 8 weeks of mTOR inhibitor therapy (either sirolimus or everolimus).

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects
2. ≥ 18 years of age
3. Diagnosis of LAM via either a. Histopathologic diagnosis b. Compatible CT chest and one of the following i. Tuberous Sclerosis Complex* ii. Angiomyolipoma or lymphangioma iii. Chylous Effusion iv. Serum VEGF-D level >800 pg/mL

   * The diagnosis of TSC will be based on the presence of at least two major criteria or one major and one or more minor features per published guidelines.(30)

Exclusion Criteria:

1. Patients with any known intrathoracic cancer (primary lung cancer or metastatic disease) or undergoing active treatment for malignancy
2. Patients with use of investigational therapies for LAM either currently or in the prior 3 months
3. Patients with body weight ≥400 pounds or body habitus or disability that will not permit the imaging protocol to be performed
4. Patients known to be pregnant or breastfeeding
5. Patients with clinically active known or suspected pulmonary infection of any type
6. Patients known or suspected to have any inborn error of metabolism
7. Patients with known type I diabetes mellitus
8. Patients who cannot have a peripheral IV for any reason
9. Patients who cannot lie flat for the duration of the PET scan
10. Patients who are claustrophobic
11. Patients with a prior allergy to contrast agents or to PET tracers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because LAM is a disease that occurs essentially only in females, the study population will consist of only females.
Enrollment: 5 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the uptake of the PET tracer throughout the entire lung and any associated neoplasms (AML, Lymphangiomas) in patients with LAM | 8 weeks
  While these imaging techniques have not been used in normal populations, the pulmonary uptake of patients with known intraabdominal malignancy will serve as control for evaluation of any potential uptake. When comparing treatment effects, each patient can serve as their own control as they will have already had imaging completed prior to the initiation of therapy. VEGF-D levels will be collected from clinical laboratory assessment or will be collected at time of enrollment, and relative elevation of VEGF-D will be compared to the relative uptake of tracer within the pulmonary parenchyma of each individual patient.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Blackwell, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No